CLINICAL TRIAL: NCT02078830
Title: EXTERNAL VENTRICULAR DRAIN ASSOCIATED INFECTIONS STUDY (EVDAI-STUDY) - A Prospective Randomised Microbiological Study for Use of 3M™ Tegaderm™ Chlorhexidinegluconate Dressing at Entry Site of EVD's to Reduce EVD-associated Infections
Brief Title: Prospective Randomised Study for Use of CHG Dressing at Entry Site of EVD's to Reduce EVD-associated Infections
Acronym: EVDAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USB-2013-024
Record Dates: First submitted 2013-11-21; First posted 2014-03-05 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Wound Contamination
Keywords: Wound Contamination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3M™ Tegaderm™ I.V. Advanced Dressing (Placebo Comparator): Placebo Dressing with the same shape like the CHG-Dressing without CHG.
  Interventions: Device: Placebo Comparator: 3M™ Tegaderm™ I.V. Advanced Dressing
- 3M™ Tegaderm™ CHG Securement Dressing (Experimental): - CHG activity at EVD entry site
  Interventions: Device: 3M™ Tegaderm™ CHG I.V. Securement Dressing

INTERVENTIONS:
Device: 3M™ Tegaderm™ CHG I.V. Securement Dressing — Chlorhexidine gluconate (CHG) has been dissolved into a soft gel pad (3x4 cm) to provide a reservoir for consistent and continuous antimicrobial action over time. The gel pad is active on contact without requiring additional moisture. CHG migrates under the catheter to provide continuous circumferential antimicrobial protection at the insertion site. Soft and conformable, the gel pad moulds around the catheter and hub.
  Arms: 3M™ Tegaderm™ CHG Securement Dressing
Device: Placebo Comparator: 3M™ Tegaderm™ I.V. Advanced Dressing — Placebo Dressing with the same shape like the CHG-Dressing without CHG.
  Arms: 3M™ Tegaderm™ I.V. Advanced Dressing

SUMMARY:
The objective of this study is to assess the efficacy of 3M™ Tegaderm™ CHG I.V. Securement Dressing at the entry-site of a EVD in reducing quantity of microorganisms (CFU/cm2) after a time period of 5 days as a surrogate marker for EVD-associated infections [1, 2], compared to a nonantimicrobial polyurethane 3M Tegaderm™ Transparent Film Dressing. We aim to investigate, if the adjunct of an additional CHG-impregnated device on a routinely basis for the daily care is as a valuable and effective option to reduce contamination of the EVD entry-site and consecutive colonization of the catheter.

DETAILED DESCRIPTION:
Randomised, parallel group, single-centre Phase IV trial comparing the change in the quantity of microorganisms (CFU/cm2) after a time period of 5 days (primary endpoint) as surrogate marker for EVD-associated infections [1, 2], in patients undergoing EVD with dressing at the entry site with 3M™ Tegaderm™ CHG I.V. Securement Dressing (study arm) versus 3M™ Tegaderm™ I.V. Advanced Dressing (standard arm). Secondary objectives are the comparison of regrowth (CFU/cm2) every 5th day before routine change of the device, cerebrospinal fluid (CSF) cultures every 2nd day and sonication of the catheter tip after explantation (secondary endpoints).

We hypothesize that bacterial contamination (CFU/cm2) of the EVD entry-site after 5 days compared to baseline (bacterial regrowth since baseline) in subjects treated with the 3M™ Tegaderm™ CHG I.V. Securement Dressing is significantly lower compared to subjects treated with 3M™ Tegaderm™ I.V. Advanced Dressing. Quantitative microbiology of the catheter tip (sonication) might be reduced by this external intervention, as well as CSF cultures.

We will use an internal pilot study design [3]. The three step procedure includes:

* initial sample size calculation
* sample size review
* final analysis.

ELIGIBILITY:
Inclusion Criteria:

- Patients following the criteria cited below are included: Patients undergoing implantation of an external ventricular drain (EVD), frontal or occipital, due to a given underlying pathology.

* Written informed consent (IC) by patients and/or independent physician [according 5.1]
* Age ≥ 18 years

Exclusion Criteria:

* Patients presenting one of the criteria cited below are excluded:
* Presence of clinical signs or laboratory findings suspicious infection
* Presence of antibiotic intake
* Traumatic Brain Injury (TBI) with evident or suspected dural breach (including skull base)
* Decision for Rifampin impregnated ventricular catheter (Bactiseal©)
* Known hypersensitivity to chlorhexidine (people from Japanese origin)
* Age < 18 years
* Participation in another study involving External Ventricular Drains
* Pregnancy or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
difference in bacterial contamination (CFU/cm2) of the EVD entry-site after 5 days as compared to baseline (CountTact™ skin sample III) | Day 5
  This colonization is proven to be the main source for catheter related infections.

SECONDARY OUTCOMES:
EVD-associated infection | day 1-X (Explantation)
  The secondary Endpoint is:
  • EVD-associated infection [according 4.3.3] is defined through a mandatory combination of:
  * Presence of bacteria at additional timepoints and from additional sampling:
  * culture from CSF every 2nd day until EVD-explantation
  * sonication of distal 4.5 cm (tip) and subsequent 5 cm (tunneled) EVD- part after explantation on day x
  * clinical signs as fever, meningism, Glasgow Coma Scale (GCS)-drop and blood signs of infection

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Mariani, MD, Study Director — Klinik und Poliklinik Neurochirurgie, Spitalstrasse 21, CH-4031 Basel; Michel Roethlisberger, MD, Principal Investigator — Klinik und Poliklinik Neurochirurgie, Spitalstrasse 21, CH-4031 Basel
Locations (1):
- Universitätsspital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Roethlisberger M, Moffa G, Fisch U, Wiggli B, Schoen S, Kelly C, Leu S, Croci D, Zumofen DW, Cueni N, Nogarth D, Schulz M, Bucher HC, Weisser-Rohacek M, Wasner MG, Widmer AF, Mariani L. Effectiveness of a Chlorhexidine Dressing on Silver-coated External Ventricular Drain-associated Colonization and Infection: A Prospective Single-blinded Randomized Controlled Clinical Trial. Clin Infect Dis. 2018 Nov 28;67(12):1868-1877. doi: 10.1093/cid/ciy393. PMID 29733329